CLINICAL TRIAL: NCT03664635
Title: A Phase I/II Safety, Dose Finding and Feasibility Trial of MB-CART20.1 in Patients with Relapsed or Resistant CD20 Positive B-NHL
Brief Title: MB-CART20.1 Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-2016-312
Record Dates: First submitted 2018-09-03; First posted 2018-09-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; B-cell Lymphoma Refractory; B-cell Lymphoma Recurrent
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I - Safety Dose Level (Experimental): In phase I three (3) + 3 patients will be treated with 1x10^5 MB-CART20.1 cells per kg body weight administered intravenously as single dose in the preceding safety dose level
  Interventions: Biological: MB-CART20.1
- Phase I - Dose Level 1 (Experimental): In phase I six (6) + 3 patients will be treated with 1x10^6 MB-CART20.1 cells per kg body weight administered intravenously as single dose in the dose level 1
  Interventions: Biological: MB-CART20.1
- Phase I - Dose Level 2 (Experimental): In phase I six (6) + 3 patients will be treated with 3x10^6 MB-CART20.1 cells per kg body weight administered intravenously as single dose in the dose level 2
  Interventions: Biological: MB-CART20.1
- Phase II (Experimental): The number of additional patients who will be treated with MB-CART20.1 cells in Phase II is depending on the number of evaluable patients treated with the maximum tolerated dose (MTD) level and the results in Part I
  Interventions: Biological: MB-CART20.1

INTERVENTIONS:
Biological: MB-CART20.1 — MB-CART20.1 consists of autologous CD20 Chimeric Antigen Receptor (CAR) transduced CD4 /CD8 enriched T cells targeting CD20-positive tumor cells in NHL
  Other Names: CD20-targeting CAR T Cells; Anti-CD20 CAR T cells

SUMMARY:
This trial is a phase I/II trial to assess safety, dose finding and feasibility of ex vivo generated MB-CART20.1 cells in patients with relapsed or refractory CD20 positive B-NHL.

DETAILED DESCRIPTION:
MB-CART20.1 consists of autologous Anti-CD20 Chimeric Antigen Receptor (CAR) transduced CD4 /CD8 enriched T cells targeting CD20-positive tumor cells in Non-Hodgkin-Lymphoma (NHL)

ELIGIBILITY:
Inclusion Criteria:

* Refractory/relapsed CD20+ B-NHL (including malignant transformation like Richter's transformation) with no curative treatment option.
* At least 18 years of age
* Estimated life expectancy of more than 3 months
* ECOG performance status (Eastern cooperative oncology group) of 0-2
* Negative serological HBV (Hepatitis B virus) test, negative testing of HCVAb (Hepatitis C virus Antibody), negative HIV1/2 (Human immunodeficiency virus 1/2 ) test within 6 weeks prior to enrollment
* No childbearing potential or negative pregnancy test at screening and before chemotherapy in women with childbearing potential.
* Signed and dated informed consent before conduct of any trial-specific procedure

Exclusion Criteria:

* Participation in another interventional trial that could interact with this trial
* Any evidence 0f CNS (Central nervous system) involvement
* Known history or presence of clinically relevant CNS pathology
* Patients with history of primary immunodeficiency,
* Patients with any history of auto-immune induced condition such as those caused by checkpoint inhibitors, MEK inhibitors or BRAF inhibitors, for example pituitary hypophysitis must be excluded
* Patients with Chronic Lymphocytic Leukemia unless suffering from malignant transformation
* Active systemic fungal, viral or bacterial infection
* Serious cardiac functional incapacity (class III or IV as defined by the New York Heart Association Classification)
* Severe pulmonary disease (DLCO (Transfer factor of the lung for carbon monoxide) and/or FEV1 (Forced expiratory volume in 1 second) < 65%, dyspnea at rest)
* Liver dysfunction as indicated by a total bilirubin, AST (Aspartate Aminotransferase), and ALT (Alanine aminotransferase) ≥ 2 the institutional ULN (Upper limit of normal) value, unless directly attributable to the patient's tumor
* Creatinine clearance <50 ml/min calculated according to the modified formula of Cockcroft and Gault
* Pregnant or lactating women
* Active secondary malignancy requiring treatment (except basal cell carcinoma or malignant tumor curatively treated by surgery) within the last 5 years before enrollment.
* Medical condition requiring prolonged use of systemic corticosteroids (> 1 month)
* Prior therapy with genetically modified substances
* Use of anti-CD20 antibodies within 4 weeks before leukapheresis
* Chemotherapy within 4 weeks prior to leukapheresis
* Other treatment within 4 weeks or two half-lives, whichever is longer before MB-CART20.1 infusion. This pertains to immunomodulatory therapies such as checkpoint inhibitors because of the influence on the immune system
* Concurrent systemic radiotherapy
* Hypersensitivity against any drug or its ingredients/impurities that is scheduled or likely to be given during trial participation e.g. as part of the mandatory lymphodepletion protocol, pre-medication for infusion, rescue medication/salvage therapies for treatment of related toxicities
* Patients in which such medication is contraindicated for other reasons than hypersensitivity (e.g. live vaccines and fludarabine)
* Patients in which trial related procedures are contraindicated as judged by the investigator, e.g. lumbar punctures for CSF (Cerebrospinal fluid) sampling
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequence of the trial and to formulate his/her own wishes correspondingly
* Patients who have a relationship of dependence or employer employee relationship to the sponsor or the investigator
* Committal to an institution on judicial or official order
* Cerebral dysfunction, legal incapacity
* Other investigational treatment within 4 weeks before IMP (Investigational Medicinal Product) infusion
* Clinically relevant autoimmune diseases or history of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Phase I - Determination of the maximum tolerated dose (MTD) | until day 28 after infusion of MB-CART20.1
  MTD is defined as the highest dose level at which < 33% of patients experience Dose Limiting Toxicity (DLT). Safety and toxicity assessment of MB-CART20.1 per adverse events (AE) reporting classified according to CTCAE version 5.0.
Phase II - Best overall response rate | 3 months after infusion of MB-CART20.1
  Response (Complete response (CR), Partial response (PR), Stable disease (SD), Progressive disease (PD)) is defined according to Cheson criteria.

SECONDARY OUTCOMES:
Phase I - Related safety and toxicity of MB-CART20.1 | months 3, 6, 9 and 12 after infusion of MB-CART20.1
  Per adverse events (AE) reporting classified according to CTCAE version 5.0.
Phase I - Best overall response rate over 4 weeks and 3 months | 4 weeks and 3 months after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase I - Best overall response rate over 1 year | 1 year after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase I - Occurrence of B-cell aplasia | 1 year after infusion of MB-CART20.1
  Circulating B cell numbers in the peripheral blood will be assessed by Flow cytometry.
Phase I - Phenotype and Persistence of MB-CART20.1 | 1 year after infusion of MB-CART20.1
  Blood samples for determination of persistence/phenotyping of infused MB-CART20.1 will be analysed.
Phase II - Best overall response rate over 1 year | 1 year after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase II - Overall response rate over 4 weeks and 3 months | 4 weeks and 3 months after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase II - Overall response rate over 1 year | 1 year after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase II - Number of patients with CR, PR, SD and PD | 1 year after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase II -Percentage of patients with CR, PR, SD and PD | 1 year after infusion of MB-CART20.1
  Response (CR, PR, SD and PD) is defined according to Cheson criteria.
Phase II - Safety and toxicity assessment of MB-CART20.1 | 1 year after infusion of MB-CART20.1
  Per adverse events (AE) reporting classified according to CTCAE version 5.0.
Phase II - Occurrence of B-cell aplasia | 1 year after infusion of MB-CART20.1
  Circulating B cell numbers in the peripheral blood will be assessed by Flow cytometry.
Phase II - Phenotype and Persistence of MB-CART20.1 | 1 year after infusion of MB-CART20.1
  Blood samples for determination of persistence/phenotyping of infused MB-CART20.1 will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof. Dr., Principal Investigator — Universitätsklinikum Köln
Locations (2):
- Germany (2):
  - University Hospital of Cologne - Clinic for Internal Medicine I, Cologne
  - Universitätsklikum Leipzig, AöR, Leipzig

IPD SHARING:
Plan to Share IPD: No